CLINICAL TRIAL: NCT01247974
Title: Prospective, Randomized Evaluation of New Onset Postoperative Atrial Fibrillation in Subjects Receiving the CorMatrix® ECM® for Pericardial Closure
Brief Title: Evaluation Of New Onset Postoperative Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-PR-1006
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation New Onset
Keywords: Coronary Artery Bypass Grafting; New Onset Postoperative Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CorMatrix ECM for Pericardial Closure (Experimental): Pericardial closure with CorMatrix ECM
  Interventions: Device: CorMatrix ECM for Pericardial Closure
- Control (No Intervention): No Pericardial Closure

INTERVENTIONS:
Device: CorMatrix ECM for Pericardial Closure — Circumferential closure of the pericardium following CABG surgery using the CorMatrix ECM for Pericardial Closure
  Arms: CorMatrix ECM for Pericardial Closure

SUMMARY:
This is a multi-center, prospective, randomized and controlled clinical trial comparing the safety and efficacy of the CorMatrix ECM for Pericardial Closure to reduce the incidence of new onset postoperative atrial fibrillation by circumferentially reconstructing the normal pericardial anatomy following isolated, first-time, CABG procedures compared to subjects that do not undergo pericardial closure. This trial will be conducted at up to 20 clinical sites in the U.S.

DETAILED DESCRIPTION:
The objective of this prospective clinical trial is to demonstrate the safety and efficacy of the CorMatrix ECM for Pericardial Closure to reduce the incidence of new onset postoperative atrial fibrillation by circumferentially reconstructing the normal pericardial anatomy following isolated, first-time, coronary artery bypass grafting (CABG) procedures as compared to subjects who did not undergo pericardial closure. Safety will be established by demonstrating that the composite clinical event rate for the ECM treatment group is not worse than the control group that did not undergo pericardial closure. The efficacy will be established by demonstrating a reduced incidence of new onset postoperative atrial fibrillation in the ECM treatment group as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 years of age or older
* This cardiac operation is the subject's first or primary cardiac operation
* The subject must be undergoing an isolated CABG procedure using a median sternotomy approach
* The subject must possess the ability to provide written Informed Consent
* The subject must express a willingness to fulfill all of the expected requirements of this clinical protocol

Exclusion Criteria:

* Prior history of atrial fibrillation
* Prior history of open heart surgery
* Prior history of pericarditis
* Prior history of anti-arrhythmia drug treatment (e.g., amiodarone, dronedarone or sotalol) in the past six months
* The subject has an implantable cardiac device (i.e., cardiac resynchronization therapy devices with and without defibrillator capabilities (CRTs and CRT-Ds), implantable cardioverter-defibrillators (ICD) and pacemakers)
* Concomitant procedure planned
* In the investigator's opinion, the subject may require prophylactic treatment with anti-arrhythmia drugs or temporary pacing postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gerdisch, M.D., Principal Investigator — St. Francis Heart Center
Locations (16):
- United States (16):
  - Trinity Medical Center, Birmingham, Alabama
  - Southeast Alabama Medical Center, Dothan, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Hospital, Mobile, Alabama
  - Saint Agnes Medical Center, Fresno, California
  - Stanford University School of Medicine, Stanford, California
  - St. Vincent's Hospital, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Saint Francis Heart Center, Indianapolis, Indiana
  - St. Luke's Hospital, Kansas City, Missouri
  - Columbia University Medical Center, New York, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Swedish Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject, Subject 011-006, was randomized in error to the ECM treatment group, but did not provide informed consent. This deviation was discovered prior to the surgery.
Groups:
- CorMatrix® ECM®: CorMatrix® ECM® for Pericardial Closure: Circumferential closure of the pericardium following CABG surgery using the CorMatrix ECM for Pericardial Closure
- Control: Pericardium is not closed
Period: Overall Study
Arm/Group | CorMatrix® ECM® | Control
Started | 217 | 222
Completed | 191 | 203
Not Completed | 26 | 19

BASELINE CHARACTERISTICS:
Groups:
- Control: No closure of pericardium
- Total: Total of all reporting groups
Arm/Group | CorMatrix® ECM® | Control | Total
Number analyzed (Participants) | 217 | 222 | 439
Age, Customized [Number; unit: participants]
  18Y and older | 217 | 222 | 439
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 104
  Male | 166 | 169 | 335
Region of Enrollment [Number; unit: participants]
  United States | 217 | 222 | 439

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint
Description: A composite endpoint consisting of the following procedure- related serious adverse events occurring within 30 days postprocedure:
  * Death
  * Myocardial Infarction (MI)
  * Stroke
  * Mediastinal Reoperation
  * Percutaneous Coronary Intervention (PCI)
Time Frame: 30 days postprocedure
Population: Performed with the FAS population using multiple imputation methods to impute values for missing or incomplete data. FAS population was defined as subjects in the ITT population who had CABG surgery and received their assigned treatment.
Measure: Number; unit: percentage of participants
Arm/Group | CorMatrix ECM for Pericardial Closure | Control
Number analyzed (Participants) | 217 | 222
percentage of participants | 3.9 | 3.6

2. Primary Outcome: Primary Effectiveness Endpoint
Description: Rate of new onset postoperative atrial fibrillation during the first seven days postoperatively or prior to hospital discharge, whichever was sooner.
Time Frame: 7 days postoperatively or hospital discharge, whichever is sooner
Population: Primary analysis was based upon the ITT population using multiple imputation to impute missing values. The ITT population was defined as all subjects who provided informed consent and were randomized in the trial.
Measure: Number; unit: percentage of participants
Arm/Group | CorMatrix ECM for Pericardial Closure | Control
Number analyzed (Participants) | 217 | 222
percentage of participants | 40.0 | 35.9

ADVERSE EVENTS:
Time Frame: 2 years
Description: The adverse events are summarized using the Full Analysis Set population, which includes 428 subjects (208 subjects in the ECM group and 220 subjects in the control group. AEs were only collected from the treated population.
Groups:
- CorMatrix ECM: CorMatrix ECM for Pericardial Closure
Arm/Group | CorMatrix ECM | Control
Serious Adverse Events (participants affected / at risk) | 76/208 | 54/220
Other Adverse Events (participants affected / at risk) | 190/208 | 189/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CorMatrix ECM (N=208) | Control (N=220)
Atrial fibrillation (Cardiac disorders) | 12 | 11
Angina pectoris (Cardiac disorders) | 10 | 6
Cardiac failure congestive (Cardiac disorders) | 7 | 6
Event led to Death (General disorders) | 7 | 10
Pneumonia (Infections and infestations) | 5 | 2
Urinary tract infection (Infections and infestations) | 3 | 3
Cerebrovascular accident (Nervous system disorders) | 3 | 4
Renal failure acute (Renal and urinary disorders) | 6 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Hypotension (Vascular disorders) | 4 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CorMatrix ECM (N=208) | Control (N=220)
Anaemia (Blood and lymphatic system disorders) | 29 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 15
Leukocytosis (Blood and lymphatic system disorders) | 9 | 7
Coagulopathy (Blood and lymphatic system disorders) | 4 | 6
Atrial Fibrillation (Cardiac disorders) | 66 | 71
Sinus Tachycardia (Cardiac disorders) | 14 | 13
Angina Pectoris (Cardiac disorders) | 18 | 8
Bradycardia (Cardiac disorders) | 8 | 13
Cardiac failure congestive (Cardiac disorders) | 11 | 9
Ventricular tachycardia (Cardiac disorders) | 8 | 7
Atrial flutter (Cardiac disorders) | 8 | 6
Sinus bradycardia (Cardiac disorders) | 3 | 10
Supraventricular tachycardia (Cardiac disorders) | 6 | 6
Cardiomegaly (Cardiac disorders) | 5 | 5
Generalised oedema (General disorders) | 12 | 10
Fatigue (General disorders) | 12 | 8
Oedema peripheral (General disorders) | 11 | 8
Asthenia (General disorders) | 5 | 6
Chest pain (General disorders) | 6 | 4
Pneumonia (Infections and infestations) | 21 | 10
Urinary tract infection (Infections and infestations) | 12 | 17
Postoperative wound infection (Infections and infestations) | 10 | 9
Bronchitis (Infections and infestations) | 8 | 7
Cellulitis (Infections and infestations) | 8 | 4
Incision site infection (Infections and infestations) | 10 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 54 | 35
Incision site pain (Injury, poisoning and procedural complications) | 11 | 8
Procedural pain (Injury, poisoning and procedural complications) | 8 | 6
Seroma (Injury, poisoning and procedural complications) | 5 | 6
Renal failure acute (Renal and urinary disorders) | 23 | 14
Urinary retention (Renal and urinary disorders) | 8 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 34 | 26
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 29 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 12 | 12
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 8
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Hypotension (Vascular disorders) | 26 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multi-site publication is not submitted within twenty-four (24) months after conclusion of the Study at all sites, Institution and/or the Principal Investigator may publish the results from Institution's site individually, subject to Sponsor's rights